CLINICAL TRIAL: NCT05262478
Title: Medium-Term Radiological And Clinical Follow-Up of Alpha-D Cervical Disk Prosthesis
Brief Title: Medium-Term Follow-Up of Alpha-D Cervical Disk Prosthesis
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet Kursat Karadag, Principal Investigator, Ataturk University
Other Study IDs: ATANEUROSURGERY-2
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Cervical Disc Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alpha-D cervical disc prosthesis: Alpha-D cervical disc prosthesis was developed jointly by the Spine Center of Koç University Faculty of Medicine and Toledo University Bioengineering Department. It was designed as a single unit to ensure user-friendly administration for surgeons, and it was designed and manufactured to reproduce the movements of the normal cervical movement segment.
  Interventions: Device: Alpha-D CDP

INTERVENTIONS:
Device: Alpha-D CDP — Alpha-D cervical disc prosthesis was developed jointly by the Spine Center of Koç University Faculty of Medicine and Toledo University Bioengineering Department. It was designed as a single unit to ensure user-friendly administration for surgeons, and it was designed and manufactured to reproduce the movements of the normal cervical movement segment.

SUMMARY:
Prostheses use subsequently became prevalent and a number of studies were conducted. However, prosthesis-associated heterotropic ossification (HO) in the segments with prostheses was reported in 2005, which disrupted mobility and caused fusion.

In the present study, we aimed to investigate the clinical outcomes, HO incidence, and prosthesis mobility in the patients following the operative use of Alpha-D disc prosthesis as developed and used by the authors to treat cervical disk diseases.

ELIGIBILITY:
Inclusion Criteria:

* cervical disc hernia
* underwent cervical discectomy and received cervical disc prostheses

Exclusion Criteria:

* history of cervical surgery,
* kyphotic deformity,
* rheumatological or other systemic diseases,
* severe osteophytes caused by advanced degenerative disc disease
* severe spinal stenosis

Ages: 27 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We included 33 patients with cervical disc hernia and associated radiculopathy upon radiological examination, who underwent a cervical discectomy and received cervical disc protheses (CDP; arthroplasty) with a single-level anterior discectomy.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Heterotropic ossification | Postoperative 18-78.months
  McAfee-Mehren classification

SECONDARY OUTCOMES:
visual analog scale | 4 and 12 months after surgery
  (0-10, 0=no pain, 10=extreme pain)
neck disability index | 4 and 12 months after surgery
  The questionnaire has 10 items concerning pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet K Karadag, Principal Investigator — Mehmet Kursat Karadag
Locations (1):
- Ataturk University, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leven D, Meaike J, Radcliff K, Qureshi S. Cervical disc replacement surgery: indications, technique, and technical pearls. Curr Rev Musculoskelet Med. 2017 Jun;10(2):160-169. doi: 10.1007/s12178-017-9398-3. PMID 28493215
- [Background] Park JH, Rhim SC, Roh SW. Mid-term follow-up of clinical and radiologic outcomes in cervical total disk replacement (Mobi-C): incidence of heterotopic ossification and risk factors. J Spinal Disord Tech. 2013 May;26(3):141-5. doi: 10.1097/BSD.0b013e31823ba071. PMID 22105106